CLINICAL TRIAL: NCT04903548
Title: Evaluating the Effects of Segmental/super Selective Treatment Utilizing Flex-dosing in Treating Unresectable HCC with Y90 SIR-Spheres
Brief Title: Evaluating the Effects of Selective Treatment Utilizing Flex-dosing for Unresectable HCC with Y90 SIR-Spheres
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 017.HEP.2020.D
Record Dates: First submitted 2020-09-22; First posted 2021-05-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirtuins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: SIRT with Y-90 resin microspheres — Selective internal radiation therapy (SIRT) with Y-90 resin microspheres (Y-90 resin SIRT) is an intra-arterial, catheter-based locoregional therapy that has been used to treat patients with unresectable HCC

SUMMARY:
The overall objective of this research study is to evaluate outcomes associated with flex-dosing in Y90 SIR-Sphere administration in a prospective cohort of unresectable HCC patients eligible for segmental/super selective treatment at Methodist Dallas Medical Center (MDMC).

DETAILED DESCRIPTION:
The overall objective of this research study is to evaluate outcomes associated with flex-dosing in Y90 SIR-Sphere administration in a prospective cohort of unresectable HCC patients eligible for segmental/super selective treatment at Methodist Dallas Medical Center (MDMC).

This study will enable physicians to be more precise in administering the correct radio-embolic dose, which will improve safety and efficacy of treatment while maintaining optimal dosing for tumor side effects. This study could potentially identify tumors earlier in the course of disease progression, which may result in more efficacious treatment and quality of life for patients. Earlier diagnosis and treatment may result in decreased costs.

This is a prospective cohort registry study. The prospective study cases will include all eligible Y90 patients, who meet the inclusion criteria who are treated beginning in May 2020 to May 2022. Follow-up of patients included in study will continue as needed in order to evaluate survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* All patients diagnosed with unresectable HCC in two of fewer hepatic segments at MDMC who undergo at least one SIRT procedure with Y-90 resin microspheres (SIR-Spheres®, Sirtex Medical Limited, Sydney, Australia) will be included in data capture. HCC is considered unresectable if it is multifocal or bilobar, or if the patient has malignant portal vein thrombosis, portal hypertension, or decompensated liver disease (Child-Pugh B or C).
* Eligible cases for inclusion are those that would have undergone Y-90 resin SIRT and had an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; platelets >60,000; creatinine <2 mg/dL; bilirubin <2 mg/dL; and international normalized ratio (INR) <1.2.

Exclusion Criteria:

* Subjects that do not meet the inclusion criteria
* Patients are not eligible for SIRT if they had any extrahepatic disease; contraindication to hepatic artery catheterization such as vascular abnormalities, bleeding diathesis, allergy to contrast dye, concurrent malignancy, refractory ascites, previous external beam radiation, or evidence of any uncorrectable flow to the gastrointestinal tract; or greater than 30 Gy of radiation estimated to be delivered to the lung based on angiography or Tc-99 microaggregated albumin scan (shunt fraction of 20% or greater).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with unresectable HCC in two of fewer hepatic segments at MDMC who undergo at least one SIRT procedure with Y-90 resin microspheres
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Patient demographics | May 2020 - 2022
  Patient demographics
Volumes for liver to be treated | May 2020 - 2022
  liver volume prior to treatment
Lobe/segment to be treated | May 2020 - 2022
  treatment location
Tumor volume | May 2020 - 2022
  volume of tumor prior to treatment
Lung Shunt | May 2020 - 2022
  Lung shunt presence
Tumor to normal ratio Tumor to Normal ratio prior to greatment | May 2020 - 2022
  T:N
Severity of liver disease | May 2020 - 2022
  Child-Pugh score
Liver synthetic function | May 2020 - 2022
  ALBI (albumin-bilirubin) score
Objective response rate | May 2020 - 2022
  using modified response evaluation criteria in solid tumors
Progression-free survival | May 2020 - 2022
  Progression-free survival
Overall survival | May 2020 - 2022
  Overall survival
Hospital-based charges/costs | May 2020 - 2022
  Hospital-based charges/costs
Liver function tests | May 2020 - 2022
  Measurement of Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline phosphatase (ALP), Albumin and total protein, Bilirubin, Prothrombin time (PT), L-lactate dehydrogenase (LD), Gamma-glutamyltransferase (GGT)
SPECT CT | May 2020 - 2022
  for missed Y90 administrations or extrahepatic Y90

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No